CLINICAL TRIAL: NCT00559494
Title: A Pilot Study to Assess Clinical Safety and Tolerance of Minocycline and Spinal Perfusion Pressure Augmentation in Acute Spinal Cord Injury
Brief Title: Minocycline and Perfusion Pressure Augmentation in Acute Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Paralyzed Veterans of America (Other); American Association of Neurological Surgeons (Other); Hotchkiss Brain Institute, University of Calgary (Other)
Responsible Party: Principal Investigator, Steve Casha, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17007; PVA2414 (Other Grant/Funding Number: Paralyzed Veterans of America)
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Spinal Cord Injuries
Keywords: complete spinal cord injury; incomplete spinal cord injury; central cord spinal cord injury; traumatic
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Minocycline; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Minocycline (Experimental)
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- SCPP augmentation (Experimental)
  Interventions: Procedure: SCPP augmentation
- SCPP control (Sham Comparator)
  Interventions: Procedure: SCPP control

INTERVENTIONS:
Drug: Minocycline — Minocycline IV BID x 7 days (first 10 patients 200 mg/dose, subsequent patients adjusted based on pharmacodynamic profiling to 800 mg loading dose, tapered 100 mg each dose to 400 mg then maintain at 400mg until day 7)
  Other Names: Minocin
  Arms: Minocycline
Drug: placebo — Normal saline 250cc via central line similar to minocycline arm administration protocol
  Other Names: control; saline
  Arms: Placebo
Procedure: SCPP augmentation — maintenance of spinal cord perfusion pressure at 75 mmHg with fluids and inotrope protocol
  Arms: SCPP augmentation
Procedure: SCPP control — maintenance of Mean arterial pressure of >65 mmHg with fluids and inotropes protocol without spinal cord perfusion pressure as target or guiding therapy
  Arms: SCPP control

SUMMARY:
While research in animal models of spinal cord injury have provided many promising insights, human studies have failed to produce effective therapies. We propose to investigate the drug Minocycline (a metalloproteinase inhibitor) for the treatment of spinal cord injured patients aiming to limit neurological injury and improve neurological outcome. This drug influences several secondary injury mechanisms implicated in spinal cord injury and has been effective in improving outcome after spinal cord injury in animal models. We also propose to examine the safety and feasibility of spinal cord perfusion pressure augmentation with a protocol of IV fluids and inotrope medications versus standard maintenance of mean arterial pressure in subjects who exhibit a decrease in perfusion pressure to less than 75 mmHg. The purpose of this pilot study is 1) to evaluate the feasibility of a clinical trial protocol for Minocycline in patients with acute spinal cord injury, and 2) to ensure adequate drug dosing and metabolic effect. After undergoing a process of informed consent, patients agreeing to participate in the study will be randomized to placebo or treatment groups in a double-blind fashion. Clinical neurological examinations, patient-reported quality of life, and functional independence categorization will be combined with serum and cerebrospinal fluid laboratory investigations to establish some of the pharmacological properties and the safety profile of this medication in this group of patients. In addition, patient tolerance to the dosing regimen will be assessed. The results of this study will provide the preliminary data necessary to plan for a larger prospective, randomized, controlled, double-blind clinical trial to assess efficacy and to further assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or over
* Motor complete or motor incomplete acute spinal cord injury involving bony spinal levels between C0 and T11
* Patient able to provide informed consent
* Randomization and commencement of administration of first drug dose within 12 hours of injury
* surgical decompression if needed to be performed within 24 hours of the injury
* subjects exhibiting spinal cord perfusion pressure (lumbar drain transduced pressure - mean arterial pressure)> 75 mmHg will be randomized to active augmentation protocol versus maintenance of mean arterial pressure

Exclusion Criteria:

* Acute spinal cord injury >12 hours old
* Isolated sensory deficit, motor intact
* Isolated cauda equina injury or injury at bony level T12 or below
* History of systemic lupus erythematosus (SLE)
* Pre-existing hepatic or renal disease
* Tetracycline hypersensitivity
* Pregnancy or breast feeding
* Isolated sensory deficit
* Isolated radicular motor deficit
* Significant leukopenia (white blood cell count < ½ times the lower limit of normal) at screening
* Elevated liver function tests (AST, ALT, alkaline phosphatase, or total bilirubin > 2 times the upper limit of normal) at screening
* Presence of systemic disease that might interfere with patient safety, compliance or evaluation of the condition under study (e.g. insulin-dependent diabetes, Lyme disease, clinically significant cardiac disease, HIV, HTLV-1)
* Associated traumatic conditions interfering with informed consent or outcome assessment (e.g. closed head injury, liver contusion)
* Known uncorrected severe coronary artery disease or evidence of active coronary ischemia (ECG changes, positive Troponin) will be excluded from SCPP randomization

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Protocol compliance, feasibility and adverse events | 2 years

SECONDARY OUTCOMES:
American Spinal Injury Association - motor score (primary clinical outcome) and sensory scores | 2 years
Short Form 36 - Quality of Life Assessment | 2 years
Functional Independence Measure | 2 years
London Handicap Scale | 2 years
Spinal Cord Injury Measure | 2 years
CSF collection (6/day) and biochemical assays | 7 days
Sequential Anatomical MRI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steven Casha, MD PhD FRCSC, Principal Investigator — University of Calgary; R. John Hurlbert, MD PhD FRCSC, Principal Investigator — University of Calgary; David Zygun, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- [Result] Casha S, Zygun D, McGowan MD, Bains I, Yong VW, Hurlbert RJ. Results of a phase II placebo-controlled randomized trial of minocycline in acute spinal cord injury. Brain. 2012 Apr;135(Pt 4):1224-36. doi: 10.1093/brain/aws072. PMID 22505632
- [Derived] Carnini A, Casha S, Yong VW, Hurlbert RJ, Braun JE. Reduction of PrP(C) in human cerebrospinal fluid after spinal cord injury. Prion. 2010 Apr-Jun;4(2):80-6. doi: 10.4161/pri.4.2.11756. Epub 2010 Apr 10. PMID 20418657